CLINICAL TRIAL: NCT00454246
Title: A Randomized, Open Label Study of the Effect of Intravenous Mircera on Hemoglobin Control in Patients Transitioning From Chronic Kidney Disease Stage 4 Through Dialysis
Brief Title: A Study of Mircera in Hemoglobin Control of Patients Transitioning to Dialysis.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision unrelated to safety or efficacy
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20337
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Results first posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; Epoetin Alfa; Darbepoetin alfa

ARMS (3):
- methoxy polyethylene glycol-epoetin beta (Experimental): 120-360 micrograms methoxy polyethylene glycol-epoetin beta subcutaneous (sc) monthly starting dose, for a minimum of 5 months to a maximum of 18 months.
  Dosage was adjusted to maintain a hemoglobin target range of ≥10 g/dL to ≤12 g/dL.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta
- Epoetin alfa (Active Comparator): Patients randomized to the reference arm continued to receive their standard of care dose and regimen of epoetin alfa subcutaneous once per week for a minimum of 5 months to a maximum of 18 months. Subcutaneous injections were to be administered in the same part of the body (ie, thigh, abdomen or arm) throughout the study.
  Dosage was adjusted to maintain a hemoglobin target range of ≥10 g/dL to ≤12 g/dL.
  Interventions: Drug: epoetin alfa
- Darbepoetin alfa (Active Comparator): Patients randomized to the reference arm continued to receive their standard of care dose and regimen of darbepoetin subcutaneous once every two weeks for a minimum of 5 months and a maximum of 18 months. Subcutaneous injections were to be administered in the same part of the body (ie, thigh, abdomen or arm) throughout the study.
  Dosage was adjusted to maintain a hemoglobin target range of ≥10 g/dL to ≤12 g/dL.
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta — Methoxy polyethylene glycol-epoetin beta was provided as a sterile single-use injectable solution in a 1-mL prefilled syringe containing 0.3 mL or 0.6 mL solution. The methoxy polyethylene glycol-epoetin beta injectable solution was formulated in sodium phosphate, sodium sulfate, mannitol, methionine and poloxamer 188, pH 6.2 and did not contain any preservative. Participants received methoxy polyethylene glycol-epoetin beta subcutaneous once a month.
  Other Names: Mircera
  Arms: methoxy polyethylene glycol-epoetin beta
Drug: epoetin alfa — Standard of care as prescribed, per individual participant, subcutaneous once per week. Subcutaneous injections were to be administered in the same part of the body (ie, thigh, abdomen or arm) throughout the study.
  Arms: Epoetin alfa
Drug: darbepoetin alfa — Standard of care as prescribed, per individual participant, darbepoetin alfa subcutaneous once every two weeks. Subcutaneous injections were to be administered in the same part of the body (ie, thigh,abdomen or arm) throughout the study.
  Arms: Darbepoetin alfa

SUMMARY:
This study will assess the efficacy and safety of methoxy polyethylene glycol-epoetin beta (Mircera) in the maintenance of hemoglobin levels in patients who have previously received treatment with epoetin alfa or darbepoetin alfa, and who are transitioning from chronic kidney disease stage 4 through dialysis. Patients will be randomized either to receive Mircera or to remain on their existing therapy; the initial monthly dose of subcutaneous (sc) Mircera (120-360 micrograms) will be based on the average weekly dose of epoetin alfa or darbepoetin alfa administered in the week preceding the switch to Mircera. At the initiation of dialysis, patients in the Mircera group will receive monthly intravenous (iv) Mircera at a starting dose based on their previous (sc) dose, and those in the control group will receive weekly (iv) epoetin alfa. The anticipated time on study treatment is 1-2 years, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic kidney disease stage IV not requiring dialysis;
* expected to initiate dialysis within 18 months;
* 15<=Glomerular Filtration Rate (GFR)<=29.

Exclusion Criteria:

* failing renal allograft in place;
* acute or chronic bleeding within 8 weeks prior to screening;
* transfusion of red blood cells within 8 weeks prior to screening;
* poorly controlled hypertension;
* immunosuppressive therapy in the 12 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (78):
- United States (78):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - El Dorado, Arkansas
  - Hot Springs, Arkansas
  - Bakersfield, California
  - Glendale, California
  - Granada Hills, California
  - Los Angeles, California
  - Orange, California
  - Palm Springs, California
  - Riverside, California
  - San Diego, California
  - Yuba City, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Stamford, Connecticut
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Beach Gardens, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Macon, Georgia
  - Meridan, Idaho
  - Evergreen Park, Illinois
  - Fort Wayne, Indiana
  - Wichita, Kansas
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Germantown, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Milwaukee, Michigan
  - Royal Oak, Michigan
  - Columbus, Mississippi
  - St Louis, Missouri
  - Omaha, Nebraska
  - Voorhees Township, New Jersey
  - West Orange, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - Flushing, New York
  - Great Neck, New York
  - Mineola, New York
  - Springfield Gardens, New York
  - Syracuse, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Maimisburg, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Lewistown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Orangeburg, South Carolina
  - Chattanooga, Tennessee
  - Dyersburg, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Alexandria, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Salem, Virginia
  - Bluefield, West Virginia
  - Morgantown, West Virginia
  - Appleton, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa | Darbepoetin Alfa
Started | 73 | 29 | 9
Completed | 0 | 0 | 0
Not Completed | 73 | 29 | 9
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Violation of selection criteria at entry | 6 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Refused Treatment | 1 | 1 | 0
Not completed — Failure to return | 1 | 0 | 0
Not completed — Early termination of study | 62 | 26 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa | Darbepoetin Alfa | Total
Number analyzed (Participants) | 69 | 26 | 9 | 104
Age Continuous [Mean (Standard Deviation); unit: years] — There were four (4) patients who did not receive at least one dose of study medication in the methoxy polyethylene glycol-epoetin beta group and three (3) in the Epoetin Alfa group.
  years | 69.8 (11.74) | 72.2 (11.48) | 69.1 (12.61) | 70.3 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 9 | 5 | 46
  Male | 37 | 17 | 4 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Able to Maintain Hemoglobin (Hb) Within 10-12 g/dL
Description: Efficacy analyses were not performed.
Time Frame: 6-7 months post initiation of dialysis
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Dose Adjustments
Description: Efficacy analyses were not performed.
Time Frame: 5 months post-randomization through onset of dialysis, and post-dialysis initiation through study end.
Measure: Number; unit: participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Assessed for AEs and SAEs
Description: The adverse events are captured in the adverse event and serious adverse event section of this database.
Time Frame: First dose of medication through 15 days post last dose (up to 8 months)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 69 | 26 | 9
participants | 69 | 26 | 9

ADVERSE EVENTS:
Time Frame: First dose of medication through 15 days post last dose (up to 8 months)
Description: The safety population is the population that received at least one dose of drug. Four patients in the methoxy polyethylene glycol-epoetin beta group and 3 patients in the Epoetin Alfa group did not receive at least one dose of drug.
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 7/69 | 4/26 | 1/9
Other Adverse Events (participants affected / at risk) | 13/69 | 7/26 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=69) | Epoetin Alfa (N=26) | Darbepoetin Alfa (N=9)
atrial flutter (Cardiac disorders) | 1 | 0 | 0
cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
catheter related infection (Infections and infestations) | 1 | 0 | 0
cellulitis (Infections and infestations) | 0 | 1 | 0
anticoagulation drug level above therapeutic (Investigations) | 1 | 0 | 0
hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
mental status changes (Psychiatric disorders) | 1 | 0 | 0
renal impairment (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=69) | Epoetin Alfa (N=26) | Darbepoetin Alfa (N=9)
urinary tract infection (Renal and urinary disorders) | 3 | 2 | 1
diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
oedema peripheral (General disorders) | 5 | 0 | 0
fatigue (General disorders) | 2 | 2 | 0
hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
nausea (Gastrointestinal disorders) | 4 | 0 | 0
skin laceration (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
dizziness (Nervous system disorders) | 1 | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
ascites (General disorders) | 0 | 0 | 1
bradycardia (Cardiac disorders) | 0 | 0 | 1
depression (Psychiatric disorders) | 0 | 0 | 1
diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights."